CLINICAL TRIAL: NCT02832076
Title: Role of Subcutaneous Negative Pressure Suction Drain Placed for Ten Days on Wound Healing in Obese Patients Undergoing Midline Laparotomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, dr mohammed elsafty, Associate Professor, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5374ASU
Record Dates: First submitted 2016-02-08; First posted 2016-07-14 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Postoperative Wound Healing

ARMS (2):
- group a (Experimental): This arm will receive subcutaneous negative suction drain for the midline wound for 10 days.
  Interventions: Procedure: Subcutaneous negative suction drain for 10 days
- group b (Active Comparator): This arm will receive closure of the midline wound without a subcutaneous drain.
  Interventions: Procedure: No subcutaneous drain

INTERVENTIONS:
Procedure: Subcutaneous negative suction drain for 10 days
  Arms: group a
Procedure: No subcutaneous drain
  Arms: group b

SUMMARY:
The aim of the study is to evaluate the role of subcutaneous negative pressure drain placed for 10 days on wound healing in female obese patients undergoing midline exploratory laparotomies for ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* BMI more than 30kg/m2
* midline laparotomies
* ovarian cancer

Exclusion Criteria:

* associated medical disorders

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-03; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
presence of a break in the skin wound | 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt